CLINICAL TRIAL: NCT02975258
Title: Adiposity and Airway Inflammation in HIV-Associated Airway Disease
Acronym: SHOP
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alison Morris, Professor, University of Pittsburgh
Other Study IDs: PRO15070529; 1R56HL128134-01A1 (NIH)
Record Dates: First submitted 2016-11-01; First posted 2016-11-29 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Asthma; HIV; Adiposity
Keywords: HIV; Asthma; Adiposity; Lung disease; Weight; Fat; Obese
MeSH Terms: conditions — Asthma; Obesity; Lung Diseases; Body Weight; Platelet Glycoprotein IV Deficiency | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, bronchial wash and cells
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Blood draw — Blood will be drawn for plasma, serum, and peripheral blood mononuclear cells.
Other: Questionnaires — The following questionnaires are administered to participants by study personnel: Gingo Asthma Questionnaire (GAQ) and the Asthma Quality of Life questionnaire (AQL).
Procedure: Spirometry — Spirometry is a simple breathing test that measures the amount of air in one's lungs and how well one can move that air by forcefully blowing 3 or more times into a mouthpiece. A series of these maneuvers will be performed under the instruction of a respiratory technician or respiratory therapist.
  Other Names: Lung function testing
Procedure: Methacholine challenge test — A methacholine challenge is a common test often used to support a diagnosis of asthma. The test consists of inhaling increasing doses of methacholine through a nebulizer to assess how quickly the participant's airways narrow.
  Other Names: Asthma Test
Radiation: Quantitative CT scans — There will be a standard chest CT and an abdominal CT. The CT scans capture contiguous volume scans acquired at slice thicknesses of 5.0 mm in the axial plane and reconstructed with 512 x 512 pixel matrices. CT examinations will encompass the entire thorax and the abdomen and will be performed during a breath-hold at end-inspiration. The investigators will measure % of lung tissue below a threshold for emphysema (i.e. -950 Hounsfield units). Measurements have been histologically-verified and give reproducible measurements. The data set is assembled and analyzed with the image data anonymized. If the participant has had a research chest CT scan done recently, only the abdomen CT will be done.
  Other Names: CT scan of the chest; CT scan of the abdomen
Procedure: Urine pregnancy test — All female participants with childbearing potential will be asked to provide a urine sample for pregnancy testing. The result of the pregnancy test must be negative in order for her to be in this research study.
Procedure: Adipose biopsy — The doctor will obtain a sample of fat cells from the participant's abdomen. Numbing medicine will be applied. A needle is placed through the skin & into the fat pad under the skin. A blunt-tip hollow cannula is then used to aspirate fat tissue through the incision.
  Other Names: Fat pad biopsy; Fat biopsy
Procedure: Exhaled nitric oxide measurement — The investigators will measure concentrations of exhaled nitric oxide by asking the participant to inhale deeply, and then exhale very slowly into a mouthpiece for between 10-15 seconds.
  Other Names: ENO measurement

SUMMARY:
The goals of this study are to 1) examine the relationships among inflammation, obesity, and asthma in people with HIV and 2) to test if special subtypes of cells or markers are present in the blood and lungs of people with HIV with asthma compared to those without asthma.

DETAILED DESCRIPTION:
The proposed study involves the recruitment of participant population and the use of data from the existing research study cohorts that have been recruited and have provided informed consent for participation. Participants meet all inclusion/exclusion criteria will be enrolled into the study. Participants in the existing research study cohorts have pulmonary function testing, chest CT scans, and blood draws at each study visit which occurs every 18 months for 3 visits. Some of the study procedures may not be repeated if they were done as part of other research projects.

1. Main study visit

   The following research procedures may be performed over the course of one or more visits to accommodate scheduling needs. The study visit will take place at the Montefiore Clinical and Translational Research Center and the University of Pittsburgh Asthma Institute in the University of Pittsburgh Medical Center - Montefiore Hospital and may take up to 4 hours to complete.
   * Informed consent
   * Medical history review and demographics
   * Review of inclusion/exclusion criteria
   * Physical examination to include vital signs, weight and height, waist, hip, and thigh circumferences.
   * Urine pregnancy test for female of childbearing potential
   * Asthma-focused and quality of life questionnaire
   * Exhaled Nitric Oxide (eNO) measurement
   * Spirometry
   * Methacholine challenge testing - will not need to be repeated if the participant had done this as part of another study in the past 6 months.
   * Chest/Abdominal CT scans (If the participant has had the Chest CT scan done within 6 months as part of other research study, they will not be repeated for study purposes. Only the Abdominal CT will be performed)
   * Research blood sampling for biomarker analyses - some of this blood will also be used for pre-bronchoscopy testing in the case that the participant qualifies and is interested in undergoing part 2, the bronchoscopy visit.
   * Adipose tissue biopsy (Fat Biopsy): performed on participants with a BMI≥25). This will be repeated if done previously because testing to be done on the fat will be different than what had been tested on the fat previously.
2. Optional sub-study

On a separate visit, only a subset of 60 selected participants will be asked to undergo the following procedures to obtain additional lung biological samples. This visit is optional for participants who are willing to participate in the bronchoscopy portion. The investigators will try to recruit an equal number (n=15 per group) of obese asthmatics, obese non-asthmatics, non-obese asthmatics, and non-obese non-asthmatics. The visit will take place in the Montefiore Clinical Translational Research Center (MUH-CTRC). The bronchoscopy procedure will take about 30-45 minutes, but the preparation and recovery time will usually make the visit about 4-8 hours total.

Participants will be expected to fast for 8 hours prior to the bronchoscopy procedure and refrain from drinking any liquids the day of the procedure. Participants may take their usual medicines with sips of water.

• Clinical laboratory testing to include complete blood count/differential/platelet count, prothrombin time/partial thromboplastin time, international Normalized Ratio, blood urea nitrogen, and creatinine prior to bronchoscopy. If the patient refuses the first blood draw, the sample is inadequate, or the labs were run more than 30 days prior to the bronchoscopy visit, a second blood sample of up to 1 tablespoon may be drawn prior to the bronchoscopy procedure to ensure the patient is healthy enough for the procedure.

If Methacholine challenge was done more than 30 days prior to the visit two date, pulmonary function tests will be repeated.

* Oral Wash: participants will be asked to gargle with salt water for 1 minute and then spit into a container to provide a sample of approximately 10mls (2 teaspoons) at this study visit.
* Tongue Scraping: tongue blade or similar object will be used to scrape the participant's tongue. This sample will be used to determine what bacteria are on the participant's tongue. This procedure should only take minutes and is not painful.
* Participants will then rinse with 10cc's of Listerine. This is to assure that there are no bacteria left behind in the participant's mouth prior to the bronchoscopy.
* Bronchoscopy with bronchoalveolar lavage (BAL), endobronchial brushing and biopsy

Under local anesthesia, participants will undergo bronchoscopy with BAL for microbiologic specimens. A light intravenous anesthetic will be titrated to provide participant comfort if necessary. Vitals signs will be monitored continuously before, during, and after the procedure. This procedure consists of 3 stages.

1. Pulmonary Lavage: During pulmonary lavage, five 50 mL washes of sterile salt-water solution will be injected through the bronchoscope. Fluid will be collected with gentle suctioning for research studies.
2. Bronchial Brushing: A small brush will be introduced through the bronchoscope and gently rubbed over a very small part of the surface of the lungs. Approximately 10 brushes will be performed to collect epithelial cells.
3. Endobronchial Biopsy: While the bronchoscope is inserted, another small instrument will be passed through the bronchoscope to take small samples (biopsies) of tissue from the walls of the airways. Up to 5 samples may be taken during this procedure.

Following the bronchoscopy procedure, participants will be closely monitored in the bronchoscopy recovery area or return to the CTRC. Rarely, the participant's asthma may worsen during or after the procedure. Appropriate medical treatments or overnight observation will be provided if needed. Participants will not be allowed to drive home after the bronchoscopy. This is because the sedatives used during the procedure may decrease driving ability. The investigators will ask for the contact name and number of the person that will pick up the participant after the bronchoscopy

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Subject who have been previously determined to be HIV positive through testing

Exclusion Criteria:

1. Pregnancy or breast-feeding
2. Contraindication to pulmonary function testing (i.e. abdominal or cataract surgery within 3 months, recent myocardial infarction, etc.)
3. Heart condition such as tachycardia, angina or arrhythmias
4. Acute respiratory infection: increasing respiratory symptoms or fever (temperature >100.4°F [38°C]) within 4 weeks of study entry
5. Hospitalization within 4 weeks of study entry
6. Uncontrolled hypertension at screening visit (systolic > 160 mm Hg or diastolic > 100 mm Hg) from an average of two or more readings (participant may return for screening after blood pressure is controlled)
7. Active cancer requiring systemic chemotherapy or radiation
8. Active infection of lungs, brain, or abdomen; or intravenous drug use or alcohol use that will impair ability to complete study investigations in the opinion of the investigator
9. History of prior lung resection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV positive individuals in the Pittsburgh area
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Adverse interaction of adiposity and HIV-associated inflammation in asthma susceptibility and airway remodeling in HIV | Baseline
  The investigator will test association of adiposity (body mass index, waist circumference, computed tomography (CT)-measured visceral adiposity) with prevalence of asthma and longitudinal progression of airway obstruction. the blood and lungs of people with HIV with asthma compared to those without asthma.

SECONDARY OUTCOMES:
Correlation between leptin and asthma susceptibility in HIV. | Baseline
  Leptin, an obesity-related inflammatory marker, levels will be compared between HIV+ asthmatics and non-asthmatics and correlated with airway remodeling on endobronchial biopsy and CT.
Correlation between adiponectin, asthma susceptibility, and airway remodeling in HIV. | Baseline
  Adiponectin, an obesity-related inflammatory marker, levels will be compared between HIV+ asthmatics and non-asthmatics and correlated with airway remodeling on endobronchial biopsy and CT.
Adipose tissue-related inflammation contributes to asthma susceptibility and airway remodeling in HIV. | Baseline
  Using abdominal adipose tissue biopsies, the investigators will phenotype adipose-specific inflammatory cells and pathways and determine associations with asthma, airway remodeling, and longitudinal progression of airway obstruction.
Low L-arginine increases asthma risk and airway remodeling in HIV. | Baseline
  The investigator will measure L-arginine in serum and bronchoalveolar lavage samples to compare levels between HIV+ asthmatics and non-asthmatics and correlate L-arginine with CT and biopsy measures of airway remodeling.
Low ADMA increases asthma risk and airway remodeling in HIV. | Baseline
  The investigator will measure ADMA in serum and bronchoalveolar lavage samples to compare levels between HIV+ asthmatics and non-asthmatics and correlate ADMA with CT and biopsy measures of airway remodeling.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Morris, MD, MS, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gingo MR, Wenzel SE, Steele C, Kessinger CJ, Lucht L, Lawther T, Busch M, Hillenbrand ME, Weinman R, Slivka WA, McMahon DK, Zhang Y, Sciurba FC, Morris A. Asthma diagnosis and airway bronchodilator response in HIV-infected patients. J Allergy Clin Immunol. 2012 Mar;129(3):708-714.e8. doi: 10.1016/j.jaci.2011.11.015. Epub 2011 Dec 15. PMID 22177327
- [Background] Miranda C, Busacker A, Balzar S, Trudeau J, Wenzel SE. Distinguishing severe asthma phenotypes: role of age at onset and eosinophilic inflammation. J Allergy Clin Immunol. 2004 Jan;113(1):101-8. doi: 10.1016/j.jaci.2003.10.041. PMID 14713914
- [Background] Holguin F, Comhair SA, Hazen SL, Powers RW, Khatri SS, Bleecker ER, Busse WW, Calhoun WJ, Castro M, Fitzpatrick AM, Gaston B, Israel E, Jarjour NN, Moore WC, Peters SP, Teague WG, Chung KF, Erzurum SC, Wenzel SE. An association between L-arginine/asymmetric dimethyl arginine balance, obesity, and the age of asthma onset phenotype. Am J Respir Crit Care Med. 2013 Jan 15;187(2):153-9. doi: 10.1164/rccm.201207-1270OC. Epub 2012 Nov 29. PMID 23204252
- [Background] Gingo MR, George MP, Kessinger CJ, Lucht L, Rissler B, Weinman R, Slivka WA, McMahon DK, Wenzel SE, Sciurba FC, Morris A. Pulmonary function abnormalities in HIV-infected patients during the current antiretroviral therapy era. Am J Respir Crit Care Med. 2010 Sep 15;182(6):790-6. doi: 10.1164/rccm.200912-1858OC. Epub 2010 Jun 3. PMID 20522793
- [Background] Crothers K, Thompson BW, Burkhardt K, Morris A, Flores SC, Diaz PT, Chaisson RE, Kirk GD, Rom WN, Huang L; Lung HIV Study. HIV-associated lung infections and complications in the era of combination antiretroviral therapy. Proc Am Thorac Soc. 2011 Jun;8(3):275-81. doi: 10.1513/pats.201009-059WR. PMID 21653528
- [Background] Gingo MR, Balasubramani GK, Kingsley L, Rinaldo CR Jr, Alden CB, Detels R, Greenblatt RM, Hessol NA, Holman S, Huang L, Kleerup EC, Phair J, Sutton SH, Seaberg EC, Margolick JB, Wisniewski SR, Morris A. The impact of HAART on the respiratory complications of HIV infection: longitudinal trends in the MACS and WIHS cohorts. PLoS One. 2013;8(3):e58812. doi: 10.1371/journal.pone.0058812. Epub 2013 Mar 12. PMID 23554932
- [Background] Grubb JR, Moorman AC, Baker RK, Masur H. The changing spectrum of pulmonary disease in patients with HIV infection on antiretroviral therapy. AIDS. 2006 May 12;20(8):1095-107. doi: 10.1097/01.aids.0000226949.64600.f9. No abstract available. PMID 16691060
- [Background] Llibre JM, Falco V, Tural C, Negredo E, Pineda JA, Munoz J, Ortega E, Videla S, Sirera G, Martinez E, Miralles C, Iribarren J, Galindo MJ, Domingo P, d'Arminio-Monforte A, Miro JM, Clotet B. The changing face of HIV/AIDS in treated patients. Curr HIV Res. 2009 Jul;7(4):365-77. doi: 10.2174/157016209788680633. PMID 19601771
- [Background] Crothers K, Huang L, Goulet JL, Goetz MB, Brown ST, Rodriguez-Barradas MC, Oursler KK, Rimland D, Gibert CL, Butt AA, Justice AC. HIV infection and risk for incident pulmonary diseases in the combination antiretroviral therapy era. Am J Respir Crit Care Med. 2011 Feb 1;183(3):388-95. doi: 10.1164/rccm.201006-0836OC. Epub 2010 Sep 17. PMID 20851926
- [Background] Akinbami LJ, Moorman JE, Bailey C, Zahran HS, King M, Johnson CA, Liu X. Trends in asthma prevalence, health care use, and mortality in the United States, 2001-2010. NCHS Data Brief. 2012 May;(94):1-8. PMID 22617340
- [Background] Moorman JE, Zahran H, Truman BI, Molla MT; Centers for Disease Control and Prevention (CDC). Current asthma prevalence - United States, 2006-2008. MMWR Suppl. 2011 Jan 14;60(1):84-6. No abstract available. PMID 21430629
- [Background] Gingo MR, Balasubramani GK, Rice TB, Kingsley L, Kleerup EC, Detels R, Seaberg EC, Greenblatt RM, Holman S, Huang L, Sutton SH, Bertolet M, Morris A. Pulmonary symptoms and diagnoses are associated with HIV in the MACS and WIHS cohorts. BMC Pulm Med. 2014 Apr 30;14:75. doi: 10.1186/1471-2466-14-75. PMID 24884738
- [Background] Lehmann S, Bakke PS, Eide GE, Gulsvik A. Bronchodilator response to adrenergic beta2-agonists: relationship to symptoms in an adult community. Respir Med. 2007 Jun;101(6):1183-90. doi: 10.1016/j.rmed.2006.11.007. Epub 2006 Dec 22. PMID 17188486
- [Background] Shore SA. Obesity, airway hyperresponsiveness, and inflammation. J Appl Physiol (1985). 2010 Mar;108(3):735-43. doi: 10.1152/japplphysiol.00749.2009. Epub 2009 Oct 29. PMID 19875711
- [Background] Beuther DA, Sutherland ER. Overweight, obesity, and incident asthma: a meta-analysis of prospective epidemiologic studies. Am J Respir Crit Care Med. 2007 Apr 1;175(7):661-6. doi: 10.1164/rccm.200611-1717OC. Epub 2007 Jan 18. PMID 17234901
- [Background] Sutherland ER, Lehman EB, Teodorescu M, Wechsler ME; National Heart, Lung, and Blood Institute's Asthma Clinical Research Network. Body mass index and phenotype in subjects with mild-to-moderate persistent asthma. J Allergy Clin Immunol. 2009 Jun;123(6):1328-34.e1. doi: 10.1016/j.jaci.2009.04.005. PMID 19501235
- [Background] Dixon AE, Pratley RE, Forgione PM, Kaminsky DA, Whittaker-Leclair LA, Griffes LA, Garudathri J, Raymond D, Poynter ME, Bunn JY, Irvin CG. Effects of obesity and bariatric surgery on airway hyperresponsiveness, asthma control, and inflammation. J Allergy Clin Immunol. 2011 Sep;128(3):508-15.e1-2. doi: 10.1016/j.jaci.2011.06.009. Epub 2011 Jul 23. PMID 21782230
- [Background] Shore SA, Schwartzman IN, Mellema MS, Flynt L, Imrich A, Johnston RA. Effect of leptin on allergic airway responses in mice. J Allergy Clin Immunol. 2005 Jan;115(1):103-9. doi: 10.1016/j.jaci.2004.10.007. PMID 15637554
- [Background] Sood A, Cui X, Qualls C, Beckett WS, Gross MD, Steffes MW, Smith LJ, Jacobs DR Jr. Association between asthma and serum adiponectin concentration in women. Thorax. 2008 Oct;63(10):877-82. doi: 10.1136/thx.2007.090803. Epub 2008 Apr 4. PMID 18390629
- [Background] Sood A, Qualls C, Schuyler M, Thyagarajan B, Steffes MW, Smith LJ, Jacobs DR Jr. Low serum adiponectin predicts future risk for asthma in women. Am J Respir Crit Care Med. 2012 Jul 1;186(1):41-7. doi: 10.1164/rccm.201110-1767OC. Epub 2012 Apr 6. PMID 22492987
- [Background] Wildman RP, Kaplan R, Manson JE, Rajkovic A, Connelly SA, Mackey RH, Tinker LF, Curb JD, Eaton CB, Wassertheil-Smoller S. Body size phenotypes and inflammation in the Women's Health Initiative Observational Study. Obesity (Silver Spring). 2011 Jul;19(7):1482-91. doi: 10.1038/oby.2010.332. Epub 2011 Jan 13. PMID 21233809
- [Background] Lumeng CN, Saltiel AR. Inflammatory links between obesity and metabolic disease. J Clin Invest. 2011 Jun;121(6):2111-7. doi: 10.1172/JCI57132. Epub 2011 Jun 1. PMID 21633179
- [Background] Shoelson SE, Lee J, Goldfine AB. Inflammation and insulin resistance. J Clin Invest. 2006 Jul;116(7):1793-801. doi: 10.1172/JCI29069. PMID 16823477
- [Background] Keaney JF Jr, Larson MG, Vasan RS, Wilson PW, Lipinska I, Corey D, Massaro JM, Sutherland P, Vita JA, Benjamin EJ; Framingham Study. Obesity and systemic oxidative stress: clinical correlates of oxidative stress in the Framingham Study. Arterioscler Thromb Vasc Biol. 2003 Mar 1;23(3):434-9. doi: 10.1161/01.ATV.0000058402.34138.11. Epub 2003 Jan 30. PMID 12615693
- [Background] Fried SK, Bunkin DA, Greenberg AS. Omental and subcutaneous adipose tissues of obese subjects release interleukin-6: depot difference and regulation by glucocorticoid. J Clin Endocrinol Metab. 1998 Mar;83(3):847-50. doi: 10.1210/jcem.83.3.4660. PMID 9506738
- [Background] Hotamisligil GS, Shargill NS, Spiegelman BM. Adipose expression of tumor necrosis factor-alpha: direct role in obesity-linked insulin resistance. Science. 1993 Jan 1;259(5091):87-91. doi: 10.1126/science.7678183.
- [Background] Feinstein R, Kanety H, Papa MZ, Lunenfeld B, Karasik A. Tumor necrosis factor-alpha suppresses insulin-induced tyrosine phosphorylation of insulin receptor and its substrates. J Biol Chem. 1993 Dec 15;268(35):26055-8. PMID 8253716
- [Background] Apovian CM, Bigornia S, Mott M, Meyers MR, Ulloor J, Gagua M, McDonnell M, Hess D, Joseph L, Gokce N. Adipose macrophage infiltration is associated with insulin resistance and vascular endothelial dysfunction in obese subjects. Arterioscler Thromb Vasc Biol. 2008 Sep;28(9):1654-9. doi: 10.1161/ATVBAHA.108.170316. Epub 2008 Jun 19. PMID 18566296
- [Background] Steinberg HO, Chaker H, Leaming R, Johnson A, Brechtel G, Baron AD. Obesity/insulin resistance is associated with endothelial dysfunction. Implications for the syndrome of insulin resistance. J Clin Invest. 1996 Jun 1;97(11):2601-10. doi: 10.1172/JCI118709. PMID 8647954
- [Background] Masia M, Padilla S, Garcia N, Jarrin I, Bernal E, Lopez N, Hernandez I, Gutierrez F. Endothelial function is impaired in HIV-infected patients with lipodystrophy. Antivir Ther. 2010;15(1):101-10. doi: 10.3851/IMP1491. PMID 20167996
- [Background] Kim JA, Montagnani M, Koh KK, Quon MJ. Reciprocal relationships between insulin resistance and endothelial dysfunction: molecular and pathophysiological mechanisms. Circulation. 2006 Apr 18;113(15):1888-904. doi: 10.1161/CIRCULATIONAHA.105.563213. PMID 16618833
- [Background] Paruthi J, Gill N, Mantzoros CS. Adipokines in the HIV/HAART-associated lipodystrophy syndrome. Metabolism. 2013 Sep;62(9):1199-205. doi: 10.1016/j.metabol.2013.04.014. Epub 2013 May 24. PMID 23706880
- [Background] Tong Q, Sankale JL, Hadigan CM, Tan G, Rosenberg ES, Kanki PJ, Grinspoon SK, Hotamisligil GS. Regulation of adiponectin in human immunodeficiency virus-infected patients: relationship to body composition and metabolic indices. J Clin Endocrinol Metab. 2003 Apr;88(4):1559-64. doi: 10.1210/jc.2002-021600. PMID 12679439
- [Background] Vigouroux C, Maachi M, Nguyen TH, Coussieu C, Gharakhanian S, Funahashi T, Matsuzawa Y, Shimomura I, Rozenbaum W, Capeau J, Bastard JP. Serum adipocytokines are related to lipodystrophy and metabolic disorders in HIV-infected men under antiretroviral therapy. AIDS. 2003 Jul 4;17(10):1503-11. doi: 10.1097/00002030-200307040-00011. PMID 12824788
- [Background] Armah KA, McGinnis K, Baker J, Gibert C, Butt AA, Bryant KJ, Goetz M, Tracy R, Oursler KK, Rimland D, Crothers K, Rodriguez-Barradas M, Crystal S, Gordon A, Kraemer K, Brown S, Gerschenson M, Leaf DA, Deeks SG, Rinaldo C, Kuller LH, Justice A, Freiberg M. HIV status, burden of comorbid disease, and biomarkers of inflammation, altered coagulation, and monocyte activation. Clin Infect Dis. 2012 Jul;55(1):126-36. doi: 10.1093/cid/cis406. Epub 2012 Apr 24. PMID 22534147
- [Background] Freiberg MS, Chang CC, Kuller LH, Skanderson M, Lowy E, Kraemer KL, Butt AA, Bidwell Goetz M, Leaf D, Oursler KA, Rimland D, Rodriguez Barradas M, Brown S, Gibert C, McGinnis K, Crothers K, Sico J, Crane H, Warner A, Gottlieb S, Gottdiener J, Tracy RP, Budoff M, Watson C, Armah KA, Doebler D, Bryant K, Justice AC. HIV infection and the risk of acute myocardial infarction. JAMA Intern Med. 2013 Apr 22;173(8):614-22. doi: 10.1001/jamainternmed.2013.3728. PMID 23459863
- [Background] Freiberg MS, Chang CC, Skanderson M, McGinnis K, Kuller LH, Kraemer KL, Rimland D, Goetz MB, Butt AA, Rodriguez Barradas MC, Gibert C, Leaf D, Brown ST, Samet J, Kazis L, Bryant K, Justice AC; Veterans Aging Cohort Study. The risk of incident coronary heart disease among veterans with and without HIV and hepatitis C. Circ Cardiovasc Qual Outcomes. 2011 Jul;4(4):425-32. doi: 10.1161/CIRCOUTCOMES.110.957415. Epub 2011 Jun 28. PMID 21712519
- [Background] Justice AC, Braithwaite RS. Lessons learned from the first wave of aging with HIV. AIDS. 2012 Jul 31;26 Suppl 1(Suppl 1):S11-8. doi: 10.1097/QAD.0b013e3283558500. PMID 22781174
- [Background] Sattler FR, He J, Letendre S, Wilson C, Sanders C, Heaton R, Ellis R, Franklin D, Aldrovandi G, Marra CM, Clifford D, Morgello S, Grant I, McCutchan JA; CHARTER Group. Abdominal obesity contributes to neurocognitive impairment in HIV-infected patients with increased inflammation and immune activation. J Acquir Immune Defic Syndr. 2015 Mar 1;68(3):281-8. doi: 10.1097/QAI.0000000000000458. PMID 25469522
- [Background] Kim DJ, Westfall AO, Chamot E, Willig AL, Mugavero MJ, Ritchie C, Burkholder GA, Crane HM, Raper JL, Saag MS, Willig JH. Multimorbidity patterns in HIV-infected patients: the role of obesity in chronic disease clustering. J Acquir Immune Defic Syndr. 2012 Dec 15;61(5):600-5. doi: 10.1097/QAI.0b013e31827303d5. PMID 23023101
- [Background] Zheng B, Leader JK, McMurray JM, Park SC, Fuhrman CR, Gur D, Sciurba FC. Automated detection and quantitative assessment of pulmonary airways depicted on CT images. Med Phys. 2007 Jul;34(7):2844-52. doi: 10.1118/1.2742777. PMID 17821992
- [Background] Elias JA, Zhu Z, Chupp G, Homer RJ. Airway remodeling in asthma. J Clin Invest. 1999 Oct;104(8):1001-6. doi: 10.1172/JCI8124. No abstract available. PMID 10525034
- [Background] Aysola RS, Hoffman EA, Gierada D, Wenzel S, Cook-Granroth J, Tarsi J, Zheng J, Schechtman KB, Ramkumar TP, Cochran R, Xueping E, Christie C, Newell J, Fain S, Altes TA, Castro M. Airway remodeling measured by multidetector CT is increased in severe asthma and correlates with pathology. Chest. 2008 Dec;134(6):1183-1191. doi: 10.1378/chest.07-2779. Epub 2008 Jul 18. PMID 18641116
- [Background] Montaudon M, Lederlin M, Reich S, Begueret H, Tunon-de-Lara JM, Marthan R, Berger P, Laurent F. Bronchial measurements in patients with asthma: comparison of quantitative thin-section CT findings with those in healthy subjects and correlation with pathologic findings. Radiology. 2009 Dec;253(3):844-53. doi: 10.1148/radiol.2533090303. Epub 2009 Sep 29. PMID 19789219
- [Background] Kosciuch J, Krenke R, Gorska K, Zukowska M, Maskey-Warzechowska M, Chazan R. Airway dimensions in asthma and COPD in high resolution computed tomography: can we see the difference? Respir Care. 2013 Aug;58(8):1335-42. doi: 10.4187/respcare.02175. Epub 2013 Jan 9. PMID 23307823
- [Background] Kurashima K, Hoshi T, Takayanagi N, Takaku Y, Kagiyama N, Ohta C, Fujimura M, Sugita Y. Airway dimensions and pulmonary function in chronic obstructive pulmonary disease and bronchial asthma. Respirology. 2012 Jan;17(1):79-86. doi: 10.1111/j.1440-1843.2011.02052.x. PMID 21883679
- [Background] Wenzel SE. Asthma phenotypes: the evolution from clinical to molecular approaches. Nat Med. 2012 May 4;18(5):716-25. doi: 10.1038/nm.2678. PMID 22561835
- [Background] Woodruff PG, Modrek B, Choy DF, Jia G, Abbas AR, Ellwanger A, Koth LL, Arron JR, Fahy JV. T-helper type 2-driven inflammation defines major subphenotypes of asthma. Am J Respir Crit Care Med. 2009 Sep 1;180(5):388-95. doi: 10.1164/rccm.200903-0392OC. Epub 2009 May 29. PMID 19483109
- [Background] Haldar P, Pavord ID, Shaw DE, Berry MA, Thomas M, Brightling CE, Wardlaw AJ, Green RH. Cluster analysis and clinical asthma phenotypes. Am J Respir Crit Care Med. 2008 Aug 1;178(3):218-224. doi: 10.1164/rccm.200711-1754OC. Epub 2008 May 14. PMID 18480428
- [Background] Moore WC, Meyers DA, Wenzel SE, Teague WG, Li H, Li X, D'Agostino R Jr, Castro M, Curran-Everett D, Fitzpatrick AM, Gaston B, Jarjour NN, Sorkness R, Calhoun WJ, Chung KF, Comhair SA, Dweik RA, Israel E, Peters SP, Busse WW, Erzurum SC, Bleecker ER; National Heart, Lung, and Blood Institute's Severe Asthma Research Program. Identification of asthma phenotypes using cluster analysis in the Severe Asthma Research Program. Am J Respir Crit Care Med. 2010 Feb 15;181(4):315-23. doi: 10.1164/rccm.200906-0896OC. Epub 2009 Nov 5. PMID 19892860
- [Background] Sutherland ER, Goleva E, King TS, Lehman E, Stevens AD, Jackson LP, Stream AR, Fahy JV, Leung DY; Asthma Clinical Research Network. Cluster analysis of obesity and asthma phenotypes. PLoS One. 2012;7(5):e36631. doi: 10.1371/journal.pone.0036631. Epub 2012 May 11. PMID 22606276
- [Background] Peters-Golden M, Swern A, Bird SS, Hustad CM, Grant E, Edelman JM. Influence of body mass index on the response to asthma controller agents. Eur Respir J. 2006 Mar;27(3):495-503. doi: 10.1183/09031936.06.00077205. PMID 16507848
- [Background] Appleton SL, Adams RJ, Wilson DH, Taylor AW, Ruffin RE; North West Adelaide Health Study Team. Central obesity is associated with nonatopic but not atopic asthma in a representative population sample. J Allergy Clin Immunol. 2006 Dec;118(6):1284-91. doi: 10.1016/j.jaci.2006.08.011. Epub 2006 Nov 7. PMID 17157658
- [Background] Holguin F, Bleecker ER, Busse WW, Calhoun WJ, Castro M, Erzurum SC, Fitzpatrick AM, Gaston B, Israel E, Jarjour NN, Moore WC, Peters SP, Yonas M, Teague WG, Wenzel SE. Obesity and asthma: an association modified by age of asthma onset. J Allergy Clin Immunol. 2011 Jun;127(6):1486-93.e2. doi: 10.1016/j.jaci.2011.03.036. PMID 21624618
- [Background] Komakula S, Khatri S, Mermis J, Savill S, Haque S, Rojas M, Brown L, Teague GW, Holguin F. Body mass index is associated with reduced exhaled nitric oxide and higher exhaled 8-isoprostanes in asthmatics. Respir Res. 2007 Apr 16;8(1):32. doi: 10.1186/1465-9921-8-32. PMID 17437645
- [Background] Ueda S, Kato S, Matsuoka H, Kimoto M, Okuda S, Morimatsu M, Imaizumi T. Regulation of cytokine-induced nitric oxide synthesis by asymmetric dimethylarginine: role of dimethylarginine dimethylaminohydrolase. Circ Res. 2003 Feb 7;92(2):226-33. doi: 10.1161/01.res.0000052990.68216.ef. PMID 12574151
- [Background] Vallance P, Leone A, Calver A, Collier J, Moncada S. Endogenous dimethylarginine as an inhibitor of nitric oxide synthesis. J Cardiovasc Pharmacol. 1992;20 Suppl 12:S60-2. doi: 10.1097/00005344-199204002-00018. PMID 1282988
- [Background] Palomo I, Contreras A, Alarcon LM, Leiva E, Guzman L, Mujica V, Icaza G, Diaz N, Gonzalez DR, Moore-Carrasco R. Elevated concentration of asymmetric dimethylarginine (ADMA) in individuals with metabolic syndrome. Nitric Oxide. 2011 May 31;24(4):224-8. doi: 10.1016/j.niox.2011.03.002. Epub 2011 Mar 17. PMID 21419857
- [Background] Comhair SA, Ricci KS, Arroliga M, Lara AR, Dweik RA, Song W, Hazen SL, Bleecker ER, Busse WW, Chung KF, Gaston B, Hastie A, Hew M, Jarjour N, Moore W, Peters S, Teague WG, Wenzel SE, Erzurum SC. Correlation of systemic superoxide dismutase deficiency to airflow obstruction in asthma. Am J Respir Crit Care Med. 2005 Aug 1;172(3):306-13. doi: 10.1164/rccm.200502-180OC. Epub 2005 May 5. PMID 15883124
- [Background] Nadeem A, Raj HG, Chhabra SK. Increased oxidative stress and altered levels of antioxidants in chronic obstructive pulmonary disease. Inflammation. 2005 Feb;29(1):23-32. doi: 10.1007/s10753-006-8965-3. PMID 16502343
- [Background] Klein E, Weigel J, Buford MC, Holian A, Wells SM. Asymmetric dimethylarginine potentiates lung inflammation in a mouse model of allergic asthma. Am J Physiol Lung Cell Mol Physiol. 2010 Dec;299(6):L816-25. doi: 10.1152/ajplung.00188.2010. Epub 2010 Oct 1. PMID 20889675
- [Background] Boger RH, Bode-Boger SM, Szuba A, Tsao PS, Chan JR, Tangphao O, Blaschke TF, Cooke JP. Asymmetric dimethylarginine (ADMA): a novel risk factor for endothelial dysfunction: its role in hypercholesterolemia. Circulation. 1998 Nov 3;98(18):1842-7. doi: 10.1161/01.cir.98.18.1842. PMID 9799202
- [Background] Miyazaki H, Matsuoka H, Cooke JP, Usui M, Ueda S, Okuda S, Imaizumi T. Endogenous nitric oxide synthase inhibitor: a novel marker of atherosclerosis. Circulation. 1999 Mar 9;99(9):1141-6. doi: 10.1161/01.cir.99.9.1141. PMID 10069780
- [Background] Scott JA, North ML, Rafii M, Huang H, Pencharz P, Subbarao P, Belik J, Grasemann H. Asymmetric dimethylarginine is increased in asthma. Am J Respir Crit Care Med. 2011 Oct 1;184(7):779-85. doi: 10.1164/rccm.201011-1810OC. PMID 21719758
- [Background] Heijink I, van Oosterhout A, Kliphuis N, Jonker M, Hoffmann R, Telenga E, Klooster K, Slebos DJ, ten Hacken N, Postma D, van den Berge M. Oxidant-induced corticosteroid unresponsiveness in human bronchial epithelial cells. Thorax. 2014 Jan;69(1):5-13. doi: 10.1136/thoraxjnl-2013-203520. Epub 2013 Aug 26. PMID 23980116
- [Background] Baker JV, Neuhaus J, Duprez D, Freiberg M, Bernardino JI, Badley AD, Nixon DE, Lundgren JD, Tracy RP, Neaton JD; INSIGHT SMART Study Group. HIV replication, inflammation, and the effect of starting antiretroviral therapy on plasma asymmetric dimethylarginine, a novel marker of endothelial dysfunction. J Acquir Immune Defic Syndr. 2012 Jun 1;60(2):128-34. doi: 10.1097/QAI.0b013e318252f99f. PMID 22421746
- [Background] Kurz K, Teerlink T, Sarcletti M, Weiss G, Zangerle R, Fuchs D. Asymmetric dimethylarginine concentrations decrease in patients with HIV infection under antiretroviral therapy. Antivir Ther. 2012;17(6):1021-7. doi: 10.3851/IMP2304. Epub 2012 Aug 15. PMID 22892398
- [Background] Parikh RV, Scherzer R, Grunfeld C, Nitta EM, Leone A, Martin JN, Deeks SG, Ganz P, Hsue PY. Elevated levels of asymmetric dimethylarginine are associated with lower CD4+ count and higher viral load in HIV-infected individuals. Atherosclerosis. 2013 Jul;229(1):246-52. doi: 10.1016/j.atherosclerosis.2013.04.025. Epub 2013 Apr 30. PMID 23711612
- [Background] Kurz K, Teerlink T, Sarcletti M, Weiss G, Zangerle R, Fuchs D. Plasma concentrations of the cardiovascular risk factor asymmetric dimethylarginine (ADMA) are increased in patients with HIV-1 infection and correlate with immune activation markers. Pharmacol Res. 2009 Dec;60(6):508-14. doi: 10.1016/j.phrs.2009.07.009. Epub 2009 Aug 3. PMID 19651212
- [Background] Jang JJ, Berkheimer SB, Merchant M, Krishnaswami A. Asymmetric dimethylarginine and coronary artery calcium scores are increased in patients infected with human immunodeficiency virus. Atherosclerosis. 2011 Aug;217(2):514-7. doi: 10.1016/j.atherosclerosis.2011.03.035. Epub 2011 Apr 5. PMID 21549379
- [Background] Gingo MR, He J, Wittman C, Fuhrman C, Leader JK, Kessinger C, Lucht L, Slivka WA, Zhang Y, McMahon DK, Sciurba FC, Morris A. Contributors to diffusion impairment in HIV-infected persons. Eur Respir J. 2014 Jan;43(1):195-203. doi: 10.1183/09031936.00157712. Epub 2013 Feb 21. PMID 23429919
- [Background] Morris A, Gingo MR, George MP, Lucht L, Kessinger C, Singh V, Hillenbrand M, Busch M, McMahon D, Norris KA, Champion HC, Gladwin MT, Zhang Y, Steele C, Sciurba FC. Cardiopulmonary function in individuals with HIV infection in the antiretroviral therapy era. AIDS. 2012 Mar 27;26(6):731-40. doi: 10.1097/QAD.0b013e32835099ae. PMID 22210636
- [Background] Wenzel SE, Schwartz LB, Langmack EL, Halliday JL, Trudeau JB, Gibbs RL, Chu HW. Evidence that severe asthma can be divided pathologically into two inflammatory subtypes with distinct physiologic and clinical characteristics. Am J Respir Crit Care Med. 1999 Sep;160(3):1001-8. doi: 10.1164/ajrccm.160.3.9812110. PMID 10471631
- [Background] Wenzel SE, Wang L, Pirozzi G. Dupilumab in persistent asthma. N Engl J Med. 2013 Sep 26;369(13):1276. doi: 10.1056/NEJMc1309809. No abstract available. PMID 24066755
- [Background] Stanley TL, Falutz J, Mamputu JC, Soulban G, Potvin D, Grinspoon SK. Effects of tesamorelin on inflammatory markers in HIV patients with excess abdominal fat: relationship with visceral adipose reduction. AIDS. 2011 Jun 19;25(10):1281-8. doi: 10.1097/QAD.0b013e328347f3f1. PMID 21516030
- [Background] Stanley TL, Falutz J, Marsolais C, Morin J, Soulban G, Mamputu JC, Assaad H, Turner R, Grinspoon SK. Reduction in visceral adiposity is associated with an improved metabolic profile in HIV-infected patients receiving tesamorelin. Clin Infect Dis. 2012 Jun;54(11):1642-51. doi: 10.1093/cid/cis251. Epub 2012 Apr 10. PMID 22495074
- [Background] Stanley TL, Feldpausch MN, Oh J, Branch KL, Lee H, Torriani M, Grinspoon SK. Effect of tesamorelin on visceral fat and liver fat in HIV-infected patients with abdominal fat accumulation: a randomized clinical trial. JAMA. 2014 Jul 23-30;312(4):380-9. doi: 10.1001/jama.2014.8334. PMID 25038357
- [Background] Ochiai M, Hayashi T, Morita M, Ina K, Maeda M, Watanabe F, Morishita K. Short-term effects of L-citrulline supplementation on arterial stiffness in middle-aged men. Int J Cardiol. 2012 Mar 8;155(2):257-61. doi: 10.1016/j.ijcard.2010.10.004. Epub 2010 Nov 9. PMID 21067832
- [Background] de Gouw HW, Verbruggen MB, Twiss IM, Sterk PJ. Effect of oral L-arginine on airway hyperresponsiveness to histamine in asthma. Thorax. 1999 Nov;54(11):1033-5. doi: 10.1136/thx.54.11.1033. PMID 10525564
- [Background] Kilpelainen M, Terho EO, Helenius H, Koskenvuo M. Validation of a new questionnaire on asthma, allergic rhinitis, and conjunctivitis in young adults. Allergy. 2001 May;56(5):377-84. doi: 10.1034/j.1398-9995.2001.056005377.x. PMID 11350300
- [Background] Crapo RO, Casaburi R, Coates AL, Enright PL, Hankinson JL, Irvin CG, MacIntyre NR, McKay RT, Wanger JS, Anderson SD, Cockcroft DW, Fish JE, Sterk PJ. Guidelines for methacholine and exercise challenge testing-1999. This official statement of the American Thoracic Society was adopted by the ATS Board of Directors, July 1999. Am J Respir Crit Care Med. 2000 Jan;161(1):309-29. doi: 10.1164/ajrccm.161.1.ats11-99. No abstract available. PMID 10619836
- [Background] New NHLBI guidelines for the diagnosis and management of asthma. National Heart, Lung and Blood Institute. Lippincott Health Promot Lett. 1997 Aug;2(7):1, 8-9. No abstract available. PMID 9300898
- [Background] Zhu Z, Lee CG, Zheng T, Chupp G, Wang J, Homer RJ, Noble PW, Hamid Q, Elias JA. Airway inflammation and remodeling in asthma. Lessons from interleukin 11 and interleukin 13 transgenic mice. Am J Respir Crit Care Med. 2001 Nov 15;164(10 Pt 2):S67-70. doi: 10.1164/ajrccm.164.supplement_2.2106070. PMID 11734470
- [Background] Kaminska M, Foley S, Maghni K, Storness-Bliss C, Coxson H, Ghezzo H, Lemiere C, Olivenstein R, Ernst P, Hamid Q, Martin J. Airway remodeling in subjects with severe asthma with or without chronic persistent airflow obstruction. J Allergy Clin Immunol. 2009 Jul;124(1):45-51.e1-4. doi: 10.1016/j.jaci.2009.03.049. Epub 2009 May 29. PMID 19481790
- [Background] Lemiere C, Ernst P, Olivenstein R, Yamauchi Y, Govindaraju K, Ludwig MS, Martin JG, Hamid Q. Airway inflammation assessed by invasive and noninvasive means in severe asthma: eosinophilic and noneosinophilic phenotypes. J Allergy Clin Immunol. 2006 Nov;118(5):1033-9. doi: 10.1016/j.jaci.2006.08.003. Epub 2006 Sep 25. PMID 17088126
- [Background] Pepe C, Foley S, Shannon J, Lemiere C, Olivenstein R, Ernst P, Ludwig MS, Martin JG, Hamid Q. Differences in airway remodeling between subjects with severe and moderate asthma. J Allergy Clin Immunol. 2005 Sep;116(3):544-9. doi: 10.1016/j.jaci.2005.06.011. PMID 16159622
- [Background] Chu HW, Halliday JL, Martin RJ, Leung DY, Szefler SJ, Wenzel SE. Collagen deposition in large airways may not differentiate severe asthma from milder forms of the disease. Am J Respir Crit Care Med. 1998 Dec;158(6):1936-44. doi: 10.1164/ajrccm.158.6.9712073. PMID 9847289
- [Background] Burdo TH, Lentz MR, Autissier P, Krishnan A, Halpern E, Letendre S, Rosenberg ES, Ellis RJ, Williams KC. Soluble CD163 made by monocyte/macrophages is a novel marker of HIV activity in early and chronic infection prior to and after anti-retroviral therapy. J Infect Dis. 2011 Jul 1;204(1):154-63. doi: 10.1093/infdis/jir214. PMID 21628670
- [Background] Tippett E, Cheng WJ, Westhorpe C, Cameron PU, Brew BJ, Lewin SR, Jaworowski A, Crowe SM. Differential expression of CD163 on monocyte subsets in healthy and HIV-1 infected individuals. PLoS One. 2011;6(5):e19968. doi: 10.1371/journal.pone.0019968. Epub 2011 May 20. PMID 21625498
- [Background] McDonald B, Moyo S, Gabaitiri L, Gaseitsiwe S, Bussmann H, Koethe JR, Musonda R, Makhema J, Novitsky V, Marlink RG, Wester CW, Essex M. Persistently elevated serum interleukin-6 predicts mortality among adults receiving combination antiretroviral therapy in Botswana: results from a clinical trial. AIDS Res Hum Retroviruses. 2013 Jul;29(7):993-9. doi: 10.1089/aid.2012.0309. Epub 2013 May 9. PMID 23590237
- [Background] O'Connor KS, Osborn L, Olson L, Blumberg SJ, Frankel MR, Srinath KP, Giambo P. Design and operation of the National Asthma Survey. Vital Health Stat 1. 2008 Aug;(46):1-122. PMID 18958992
- [Background] Juniper EF, Svensson K, Mork AC, Stahl E. Measuring health-related quality of life in adults during an acute asthma exacerbation. Chest. 2004 Jan;125(1):93-7. doi: 10.1378/chest.125.1.93. PMID 14718426
- [Background] Definition and classification of chronic bronchitis for clinical and epidemiological purposes. A report to the Medical Research Council by their Committee on the Aetiology of Chronic Bronchitis. Lancet. 1965 Apr 10;1(7389):775-9. No abstract available. PMID 4165081
- [Background] Pellegrino R, Viegi G, Brusasco V, Crapo RO, Burgos F, Casaburi R, Coates A, van der Grinten CP, Gustafsson P, Hankinson J, Jensen R, Johnson DC, MacIntyre N, McKay R, Miller MR, Navajas D, Pedersen OF, Wanger J. Interpretative strategies for lung function tests. Eur Respir J. 2005 Nov;26(5):948-68. doi: 10.1183/09031936.05.00035205. No abstract available. PMID 16264058
- [Background] Wang Z, Gu S, Leader JK, Kundu S, Tedrow JR, Sciurba FC, Gur D, Siegfried JM, Pu J. Optimal threshold in CT quantification of emphysema. Eur Radiol. 2013 Apr;23(4):975-84. doi: 10.1007/s00330-012-2683-z. Epub 2012 Nov 1. PMID 23111815
- [Background] Nakano Y, Wong JC, de Jong PA, Buzatu L, Nagao T, Coxson HO, Elliott WM, Hogg JC, Pare PD. The prediction of small airway dimensions using computed tomography. Am J Respir Crit Care Med. 2005 Jan 15;171(2):142-6. doi: 10.1164/rccm.200407-874OC. Epub 2004 Oct 29. PMID 15516531
- [Background] Patel BD, Coxson HO, Pillai SG, Agusti AG, Calverley PM, Donner CF, Make BJ, Muller NL, Rennard SI, Vestbo J, Wouters EF, Hiorns MP, Nakano Y, Camp PG, Nasute Fauerbach PV, Screaton NJ, Campbell EJ, Anderson WH, Pare PD, Levy RD, Lake SL, Silverman EK, Lomas DA; International COPD Genetics Network. Airway wall thickening and emphysema show independent familial aggregation in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2008 Sep 1;178(5):500-5. doi: 10.1164/rccm.200801-059OC. Epub 2008 Jun 19. PMID 18565956
- [Background] Murphy RA, Reinders I, Register TC, Ayonayon HN, Newman AB, Satterfield S, Goodpaster BH, Simonsick EM, Kritchevsky SB, Harris TB. Associations of BMI and adipose tissue area and density with incident mobility limitation and poor performance in older adults. Am J Clin Nutr. 2014 May;99(5):1059-65. doi: 10.3945/ajcn.113.080796. Epub 2014 Feb 12. PMID 24522448
- [Background] Veraldi KL, Gibson BT, Yasuoka H, Myerburg MM, Kelly EA, Balzar S, Jarjour NN, Pilewski JM, Wenzel SE, Feghali-Bostwick CA. Role of insulin-like growth factor binding protein-3 in allergic airway remodeling. Am J Respir Crit Care Med. 2009 Oct 1;180(7):611-7. doi: 10.1164/rccm.200810-1555OC. Epub 2009 Jul 16. PMID 19608721
- [Background] Chu HW, Balzar S, Seedorf GJ, Westcott JY, Trudeau JB, Silkoff P, Wenzel SE. Transforming growth factor-beta2 induces bronchial epithelial mucin expression in asthma. Am J Pathol. 2004 Oct;165(4):1097-106. doi: 10.1016/s0002-9440(10)63371-8. PMID 15466377
- [Background] Moore WC, Evans MD, Bleecker ER, Busse WW, Calhoun WJ, Castro M, Chung KF, Erzurum SC, Curran-Everett D, Dweik RA, Gaston B, Hew M, Israel E, Mayse ML, Pascual RM, Peters SP, Silveira L, Wenzel SE, Jarjour NN; National Heart, Lung, and Blood Institute's Severe Asthma Research Group. Safety of investigative bronchoscopy in the Severe Asthma Research Program. J Allergy Clin Immunol. 2011 Aug;128(2):328-336.e3. doi: 10.1016/j.jaci.2011.02.042. Epub 2011 Apr 15. PMID 21496892
- [Background] Vanderweele TJ, Vansteelandt S. Odds ratios for mediation analysis for a dichotomous outcome. Am J Epidemiol. 2010 Dec 15;172(12):1339-48. doi: 10.1093/aje/kwq332. Epub 2010 Oct 29. PMID 21036955
- [Background] Vittinghoff E, Sen S, McCulloch CE. Sample size calculations for evaluating mediation. Stat Med. 2009 Feb 15;28(4):541-57. doi: 10.1002/sim.3491. PMID 19065627
- [Background] Poirier CD, Inhaber N, Lalonde RG, Ernst P. Prevalence of bronchial hyperresponsiveness among HIV-infected men. Am J Respir Crit Care Med. 2001 Aug 15;164(4):542-5. doi: 10.1164/ajrccm.164.4.2010019. PMID 11520712
- [Background] Weisberg SP, McCann D, Desai M, Rosenbaum M, Leibel RL, Ferrante AW Jr. Obesity is associated with macrophage accumulation in adipose tissue. J Clin Invest. 2003 Dec;112(12):1796-808. doi: 10.1172/JCI19246. PMID 14679176
- [Background] Lugogo NL, Hollingsworth JW, Howell DL, Que LG, Francisco D, Church TD, Potts-Kant EN, Ingram JL, Wang Y, Jung SH, Kraft M. Alveolar macrophages from overweight/obese subjects with asthma demonstrate a proinflammatory phenotype. Am J Respir Crit Care Med. 2012 Sep 1;186(5):404-11. doi: 10.1164/rccm.201109-1671OC. Epub 2012 Jul 5. PMID 22773729 (Retraction: PMID 26177181 Am J Respir Crit Care Med. 2015 Jul 15;192(2):264)
- [Background] Pao V, Lee GA, Grunfeld C. HIV therapy, metabolic syndrome, and cardiovascular risk. Curr Atheroscler Rep. 2008 Feb;10(1):61-70. doi: 10.1007/s11883-008-0010-6. PMID 18366987
- [Background] Cocchi F, DeVico AL, Garzino-Demo A, Arya SK, Gallo RC, Lusso P. Identification of RANTES, MIP-1 alpha, and MIP-1 beta as the major HIV-suppressive factors produced by CD8+ T cells. Science. 1995 Dec 15;270(5243):1811-5. doi: 10.1126/science.270.5243.1811. PMID 8525373
- [Background] Belda J, Leigh R, Parameswaran K, O'Byrne PM, Sears MR, Hargreave FE. Induced sputum cell counts in healthy adults. Am J Respir Crit Care Med. 2000 Feb;161(2 Pt 1):475-8. doi: 10.1164/ajrccm.161.2.9903097. PMID 10673188
- [Background] Spanevello A, Confalonieri M, Sulotto F, Romano F, Balzano G, Migliori GB, Bianchi A, Michetti G. Induced sputum cellularity. Reference values and distribution in normal volunteers. Am J Respir Crit Care Med. 2000 Sep;162(3 Pt 1):1172-4. doi: 10.1164/ajrccm.162.3.9908057. PMID 10988149
- [Background] Mallon PW, Sedwell R, Rogers G, Nolan D, Unemori P, Hoy J, Samaras K, Kelleher A, Emery S, Cooper DA, Carr A; Rosey Investigators. Effect of rosiglitazone on peroxisome proliferator-activated receptor gamma gene expression in human adipose tissue is limited by antiretroviral drug-induced mitochondrial dysfunction. J Infect Dis. 2008 Dec 15;198(12):1794-803. doi: 10.1086/593179. PMID 18954260
- [Background] Kerzerho J, Maazi H, Speak AO, Szely N, Lombardi V, Khoo B, Geryak S, Lam J, Soroosh P, Van Snick J, Akbari O. Programmed cell death ligand 2 regulates TH9 differentiation and induction of chronic airway hyperreactivity. J Allergy Clin Immunol. 2013 Apr;131(4):1048-57, 1057.e1-2. doi: 10.1016/j.jaci.2012.09.027. Epub 2012 Nov 20. PMID 23174661
- [Background] McLaughlin T, Stuhlinger M, Lamendola C, Abbasi F, Bialek J, Reaven GM, Tsao PS. Plasma asymmetric dimethylarginine concentrations are elevated in obese insulin-resistant women and fall with weight loss. J Clin Endocrinol Metab. 2006 May;91(5):1896-900. doi: 10.1210/jc.2005-1441. Epub 2006 Feb 28. PMID 16507636
- [Background] Tran CT, Leiper JM, Vallance P. The DDAH/ADMA/NOS pathway. Atheroscler Suppl. 2003 Dec;4(4):33-40. doi: 10.1016/s1567-5688(03)00032-1. PMID 14664901
- [Background] Nielsen F, Mikkelsen BB, Nielsen JB, Andersen HR, Grandjean P. Plasma malondialdehyde as biomarker for oxidative stress: reference interval and effects of life-style factors. Clin Chem. 1997 Jul;43(7):1209-14. PMID 9216458
- [Background] Maiolino G, Rossitto G, Caielli P, Bisogni V, Rossi GP, Calo LA. The role of oxidized low-density lipoproteins in atherosclerosis: the myths and the facts. Mediators Inflamm. 2013;2013:714653. doi: 10.1155/2013/714653. Epub 2013 Oct 3. PMID 24222937
- [Background] Teerlink T, Nijveldt RJ, de Jong S, van Leeuwen PA. Determination of arginine, asymmetric dimethylarginine, and symmetric dimethylarginine in human plasma and other biological samples by high-performance liquid chromatography. Anal Biochem. 2002 Apr 15;303(2):131-7. doi: 10.1006/abio.2001.5575. PMID 11950212
- [Background] Deeks SG, Lewin SR, Havlir DV. The end of AIDS: HIV infection as a chronic disease. Lancet. 2013 Nov 2;382(9903):1525-33. doi: 10.1016/S0140-6736(13)61809-7. Epub 2013 Oct 23. PMID 24152939
- [Background] Finkel T, Holbrook NJ. Oxidants, oxidative stress and the biology of ageing. Nature. 2000 Nov 9;408(6809):239-47. doi: 10.1038/35041687. PMID 11089981
- [Background] Modena BD, Tedrow JR, Milosevic J, Bleecker ER, Meyers DA, Wu W, Bar-Joseph Z, Erzurum SC, Gaston BM, Busse WW, Jarjour NN, Kaminski N, Wenzel SE. Gene expression in relation to exhaled nitric oxide identifies novel asthma phenotypes with unique biomolecular pathways. Am J Respir Crit Care Med. 2014 Dec 15;190(12):1363-72. doi: 10.1164/rccm.201406-1099OC. PMID 25338189